CLINICAL TRIAL: NCT03222609
Title: A Phase 2 Open-Label Study Evaluating Tolerability and Efficacy of Navitoclax Alone or in Combination With Ruxolitinib in Subjects With Myelofibrosis (REFINE)
Brief Title: A Study Evaluating Tolerability and Efficacy of Navitoclax Alone or in Combination With Ruxolitinib in Participants With Myelofibrosis
Acronym: REFINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16-109; 2017-001398-17 (EudraCT Number)
Expanded Access: NCT03592576 (No longer available)
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Myelofibrosis (MF)
Keywords: Post-polycythemia vera MF (PPV-MF); Post-essential thrombocythemia (PET-MF); ruxolitinib; navitoclax; splenic volume; Primary Myelofibrosis; Jakafi; enlarged spleen; splenomegaly; ABT 263; bone marrow fibrosis
MeSH Terms: conditions — Primary Myelofibrosis; Splenomegaly | interventions — ruxolitinib; navitoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Navitoclax + ruxolitinib (Cohort 1a) (Experimental): Participants must have received ruxolitinib for at least 12 weeks and on stable dose of ≥10 mg tablets orally twice daily (BID) for ≥8 weeks prior to the 1st dose of navitoclax. Navitoclax tablets are administered once daily (QD) at a starting dose of 50 mg. This was increased after approximately ≥7 days to next dose level if platelet count is ≥75 × 10^9/L up to a maximum dose of navitoclax 300 mg QD. Participants continued their treatment until the end of clinical benefit, unacceptable toxicity, or they met other protocol criteria for discontinuation (whichever occurred first).
  Interventions: Drug: Ruxolitinib; Drug: Navitoclax
- Navitoclax + ruxolitinib (Cohort 1b) (Experimental): Those receiving ruxolitinib at Screening must be on a stable dose ≥10 mg tablets orally twice daily (BID) for ≥ 4 weeks prior to 1st dose of navitoclax. Those not receiving ruxolitinib at Screening received 10 mg ruxolitinib BID starting on Day 1. Navitoclax tablets were administered orally once daily (QD) per Baseline platelet count (>150 × 10^9/L starting dose of 200 mg; ≤150 × 10^9/L starting dose of 100 mg, which could be increased to 200 mg QD after 7 days provided platelet count is ≥75 × 10^9/L). Navitoclax didn't exceed 200 mg QD for first 24 weeks of treatment. After Week 24 disease assessment, navitoclax dose was increased to 300 mg QD at discretion of the Investigator for those with suboptimal spleen response defined as failure to achieve spleen volume reduction of at least 10% per imaging. Participants continued their treatment until the end of clinical benefit, unacceptable toxicity, or they met other protocol criteria for discontinuation (whichever occurred first).
  Interventions: Drug: Ruxolitinib; Drug: Navitoclax
- Navitoclax (Cohort 2) (Experimental): Participants must have received prior treatment with a Janus Kinase 2 (JAK-2) inhibitor. Those with Baseline platelet count >150 × 10^9/L initiated navitoclax film-coated tablets orally once daily (QD) at the starting dose of 200 mg. Those with a Baseline platelet count ≤150 × 10^9/L initiated navitoclax film-coated tablets orally once daily (QD) at the starting dose of 100 mg, which could be increased to 200 mg once daily after 7 days provided the platelet count is ≥75 × 10^9/L. Navitoclax didn't exceed 200 mg QD for the first 24 weeks of treatment. After Week 24 disease assessment, navitoclax dose may be increased to 300 mg QD at discretion of the Investigator for those with suboptimal spleen response defined as failure to achieve spleen volume reduction of at least 10% per imaging. Participants continued their treatment until the end of clinical benefit, unacceptable toxicity, or they met other protocol criteria for discontinuation (whichever occurred first).
  Interventions: Drug: Navitoclax
- Navitoclax + ruxolitinib (Cohort 3) (Experimental): Prior treatment with a Janus Kinase 2 (JAK-2) or Bromodomain and Extra-Terminal motif (BET) proteins inhibitor was prohibited. Ruxolitinib tablets administered orally twice daily (BID) based on Baseline platelet count as per the local approved label. Navitoclax tablets were administered orally once daily (QD) per Baseline platelet count (>150 × 10^9/L starting dose of 200 mg; ≤150 × 10^9/L starting dose of 100 mg, which could be increased to 200 mg QD after 7 days provided platelet count is ≥75 × 10^9/L). Navitoclax didn't exceed 200 mg QD for first 24 weeks of treatment. After Week 24 disease assessment, navitoclax dose may be increased to 300 mg QD at discretion of Investigator for those with suboptimal spleen response defined as failure to achieve spleen volume reduction of at least 10% per imaging. Participants continued their treatment until the end of clinical benefit, unacceptable toxicity, or they met other protocol criteria for discontinuation (whichever occurred first).
  Interventions: Drug: Ruxolitinib; Drug: Navitoclax

INTERVENTIONS:
Drug: Ruxolitinib — Tablet; Oral
  Other Names: Jakafi
  Arms: Navitoclax + ruxolitinib (Cohort 1a); Navitoclax + ruxolitinib (Cohort 1b); Navitoclax + ruxolitinib (Cohort 3)
Drug: Navitoclax — Film-coated tablet; Oral
  Other Names: ABT-263

SUMMARY:
This is a Phase 2 open-label, multicenter study evaluating tolerability and efficacy of navitoclax alone or when added to ruxolitinib in participants with myelofibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Participants with documented diagnosis of intermediate-2 or high-risk primary Myelofibrosis, Post Polycythemia Vera Myelofibrosis or Post-essential Thrombocythemia Myelofibrosis.
* Participant must be ineligible due to age, comorbidities, or unfit for unrelated or unmatched donor transplantation or unwilling to undergo stem cell transplantation at time of study entry.
* Eastern Cooperative Oncology Group (ECOG) of 0, 1, or 2.
* Prior treatment must meet at least one of the following criteria:

  * Prior or current treatment with ruxolitinib and no prior treatment with a Bromodomain and Extra-Terminal motif (BET) proteins inhibitor or another Janus Kinase 2 (JAK-2) inhibitor, and meet all of the following criteria:

    * Ruxolitinib treatment must meet at least one of the following criteria:

      * Ruxolitinib treatment for >=24 weeks with lack of efficacy defined as a lack of spleen response (refractory) or a loss of spleen or symptom response (relapsed)
      * Ruxolitinib treatment for <24 weeks with documented disease progression on spleen measurements while on ruxolitinib as defined in the protocol:
      * Ruxolitinib treatment for >=28 days with intolerance defined as new red blood cell transfusion requirement (at least 2 units/month for 2 months) while receiving a total daily ruxolitinib dose of >=30 mg but unable to reduce dose further due to lack of efficacy.
    * If receiving ruxolitinib at the time of screening, must currently be on a stable dose >=10 mg twice daily of ruxolitinib for >=4 weeks prior to the 1st dose of navitoclax.
    * Participant has at least 2 symptoms each with a score >=3 or a total score of >=12, as measured by the Myelofibrosis Symptom Assessment Form (MFSAF) v4.0 on at least 4 out of 7 days during screening prior to study drug dosing; OR
  * Prior treatment with a JAK-2 inhibitor and meet one of the following criteria:

    * Prior treatment with a JAK-2 inhibitor for at least 12 weeks
    * Prior treatment with a JAK-2 inhibitor for >=28 days complicated by either development of red blood cell transfusion requirement (at least 2 units/month for 2 months) OR Grade >= 3 adverse events of thrombocytopenia, anemia, hematoma and/or hemorrhage while on JAK-2 inhibitor treatment; OR
  * No prior treatment with a JAK-2 or BET inhibitor.
* Participant has splenomegaly as defined in the protocol.
* Participant must meet the laboratory parameters (adequate bone marrow, renal and hepatic function) as defined in the protocol.

Exclusion Criteria:

* Splenic irradiation within 6 months prior to screening, or prior splenectomy.
* Leukemic transformation (> 10% blasts in peripheral blood or bone marrow aspirate/biopsy).
* Participant is currently on medications that interfere with coagulation (including warfarin) or platelet function within 3 days prior to the first dose of study drug or during the study treatment period with the exception of low dose aspirin (up to 100 mg/day) and low-molecular-weight heparin.
* Prior therapy with a BH3 mimetic compound or stem cell transplantation.
* Participant has received strong CYP3A inhibitors (e.g., ketoconazole, clarithromycin) or moderate CYP3A inhibitors (e.g., fluconazole) within 14 days prior to the administration of the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2025-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (91):
- United States (33):
  - UAB Comprehensive Cancer Cente /ID# 165464, Birmingham, Alabama
  - TOI Clinical Research /ID# 222546, Cerritos, California
  - City of Hope /ID# 221395, Duarte, California
  - Moores Cancer Center at UC San Diego /ID# 164084, La Jolla, California
  - Long Beach Memorial Medical Ct /ID# 230148, Long Beach, California
  - University of Southern California /ID# 164095, Los Angeles, California
  - Colorado Blood Cancer Institute /ID# 224250, Denver, Colorado
  - Baptist MD Anderson Cancer Center - Jacksonville /ID# 222548, Jacksonville, Florida
  - Mayo Clinic /ID# 164201, Jacksonville, Florida
  - Moffitt Cancer Center /ID# 164082, Tampa, Florida
  - University of Chicago Medicine /ID# 164115, Chicago, Illinois
  - Mid Illinois Hematology & Oncology Associates, Ltd /ID# 230536, Normal, Illinois
  - Indiana Blood & Marrow Transpl /ID# 165075, Indianapolis, Indiana
  - Duplicate_American Oncology Partners of Maryland, PA /ID# 231299, Bethesda, Maryland
  - Dana-Farber Cancer Institute /ID# 162675, Boston, Massachusetts
  - University of Massachusetts - Worcester /ID# 222547, Worcester, Massachusetts
  - Henry Ford Hospital /ID# 162682, Detroit, Michigan
  - Ascension Providence Southfield Cancer Center /ID# 223876, Southfield, Michigan
  - MidAmerica Division, Inc. /ID# 222058, Kansas City, Missouri
  - Weill Cornell Medical College /ID# 162679, New York, New York
  - The Ohio State University /ID# 217402, Columbus, Ohio
  - Bend Memorial Clinic /ID# 224184, Bend, Oregon
  - West Penn Hospital /ID# 222618, Pittsburgh, Pennsylvania
  - Duplicate_Medical University of South Carolina /ID# 222597, Charleston, South Carolina
  - Prairie Lakes Healthcare System /ID# 224358, Watertown, South Dakota
  - Tennessee Oncology-Nashville Centennial /ID# 221410, Nashville, Tennessee
  - Texas Oncology - West Texas /ID# 224784, Abilene, Texas
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center /ID# 225159, Dallas, Texas
  - Oncology Consultants /ID# 230930, Houston, Texas
  - MD Anderson Cancer Center at Texas Medical Center /ID# 162683, Houston, Texas
  - University of Texas Health San Antonio MD Anderson Cancer Center /ID# 164094, San Antonio, Texas
  - Utah Cancer Specialists Salt Lake Clinic /ID# 222806, Salt Lake City, Utah
  - University of Utah /ID# 164116, Salt Lake City, Utah
- Australia (5):
  - The Kinghorn Cancer Centre /ID# 214657, Darlinghurst, New South Wales
  - Barwon Health /ID# 222430, Geelong, Victoria
  - Peter MacCallum Cancer Ctr /ID# 218352, Melbourne, Victoria
  - The Alfred Hospital /ID# 215545, Melbourne, Victoria
  - Fiona Stanley Hospital /ID# 216809, Murdoch, Western Australia
- Canada (3):
  - Duplicate_University of Alberta Hospital - Division of Hematology /ID# 217698, Edmonton, Alberta
  - University Health Network_Princess Margaret Cancer Centre /ID# 214483, Toronto, Ontario
  - McGill University Health Center Research Institute /ID# 223976, Montreal, Quebec
- Croatia (4):
  - Clinical Hospital Dubrava /ID# 230504, Zagreb, City of Zagreb
  - Klinicka bolnica Merkur /ID# 230599, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 230602, Zagreb, City of Zagreb
  - Klinicki Bolnicki Centar (KBC) Split /ID# 230601, Split, Split-Dalmatia County
- Greece (2):
  - General Hospital of Athens Laiko /ID# 230394, Athens, Attica
  - Duplicate_University General Hospital Attikon /ID# 230395, Athens, Attica
- Hungary (3):
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz /ID# 230585, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Semmelweis Egyetem /ID# 230518, Budapest
  - Duplicate_Del-pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet /ID# 230306, Budapest
- Israel (4):
  - Hadassah Medical Center-Hebrew University /ID# 230310, Jerusalem, Jerusalem
  - Galilee Medical Center /ID# 230397, Nahariya, Northern District
  - Assuta Ashdod Medical Center /ID# 230396, Ashdod, Southern District
  - Tel Aviv Sourasky Medical Center /ID# 230311, Tel Aviv, Tel Aviv
- Italy (8):
  - IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 230012, Bologna, Emilia-Romagna
  - Azienda Ospedaliero Universitaria Careggi /ID# 214555, Florence, Firenze
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 214553, Rome, Roma
  - ASST Papa Giovanni XXIII /ID# 214900, Bergamo
  - ASST degli Spedali Civili di Brescia /ID# 230420, Brescia
  - AOU Policlinico G. Rodolico - San Marco /ID# 214549, Catania
  - Grande Ospedale Metropolitano Bianchi - Melacrino - Morelli P.O. Riuniti /ID# 230011, Reggio Calabria
  - ASST Sette Laghi - Ospedale Di Circolo E Fondazione Macchi Varese /ID# 214551, Varese
- Japan (10):
  - Fujita Health University Hospital /ID# 221539, Toyoake, Aichi-ken
  - Aomori Prefectural Central Hospital /ID# 221773, Aomori, Aomori
  - Kyushu University Hospital /ID# 222691, Fukuoka, Fukuoka
  - Sapporo Hokuyu Hospital /ID# 222693, Sapporo, Hokkaido
  - Kansai Medical University Hospital /ID# 222690, Hirakata-shi, Osaka
  - Kindai University Hospital /ID# 222689, Osakasayama-shi, Osaka
  - Duplicate_Dokkyo Medical University Saitama Medical Center /ID# 222332, Koshigaya-shi, Saitama
  - Juntendo University Hospital /ID# 221484, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital /ID# 222692, Bunkyo-ku, Tokyo
  - University of Yamanashi Hospital /ID# 221700, Chuo-shi, Yamanashi
- Puerto Rico (2):
  - VA Caribbean Healthcare System /ID# 222416, San Juan
  - Hospital del Centro Comprensivo de Cancer de la UPR /ID# 222544, San Juan
- South Korea (2):
  - Seoul National University Hospital /ID# 230380, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 230381, Seoul, Seoul Teugbyeolsi
- Spain (8):
  - Hospital Universitario Germans Trias i Pujol /ID# 214704, Badalona, Barcelona
  - Duplicate_CLINICA UNIVERSIDAD DE NAVARRA-Pamplona /ID# 230718, Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron /ID# 222415, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 214676, Madrid
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 230719, Madrid
  - Hospital Universitario 12 de Octubre /ID# 214710, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 214709, Málaga
  - Hospital Regional Universitario de Malaga /ID# 230858, Málaga
- Taiwan (2):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 230371, Kaohsiung City, Kaohsiung
  - National Cheng Kung University Hospital /ID# 230372, Tainan
- United Kingdom (5):
  - Guys and St Thomas NHS Foundation Trust /ID# 164110, London, Greater London
  - Oxford University Hospitals NHS Foundation Trust /ID# 214503, Oxford, Oxfordshire
  - Belfast Health and Social Care Trust /ID# 216991, Belfast
  - The Christie Hospital /ID# 164111, Manchester
  - Aneurin Bevan University Health Board /ID# 230332, Newport

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Pemmaraju N, Somervaille TCP, Palandri F, Harrison C, Komrokji RS, Perkins A, Ayala Diaz RM, Lavie D, Tomita A, Feng Y, Qin Q, Harb J, Polepally AR, Potluri J, Garcia JS. Addition of navitoclax to ruxolitinib for patients with myelofibrosis with progression or suboptimal response. Blood Neoplasia. 2024 Nov 2;2(1):100056. doi: 10.1016/j.bneo.2024.100056. eCollection 2025 Feb. PMID 40454409
- [Derived] Pemmaraju N, Garcia JS, Potluri J, Harb JG, Sun Y, Jung P, Qin QQ, Tantravahi SK, Verstovsek S, Harrison C. Addition of navitoclax to ongoing ruxolitinib treatment in patients with myelofibrosis (REFINE): a post-hoc analysis of molecular biomarkers in a phase 2 study. Lancet Haematol. 2022 Jun;9(6):e434-e444. doi: 10.1016/S2352-3026(22)00116-8. Epub 2022 May 13. PMID 35576960
- [Derived] Harrison CN, Garcia JS, Somervaille TCP, Foran JM, Verstovsek S, Jamieson C, Mesa R, Ritchie EK, Tantravahi SK, Vachhani P, O'Connell CL, Komrokji RS, Harb J, Hutti JE, Holes L, Masud AA, Nuthalapati S, Potluri J, Pemmaraju N. Addition of Navitoclax to Ongoing Ruxolitinib Therapy for Patients With Myelofibrosis With Progression or Suboptimal Response: Phase II Safety and Efficacy. J Clin Oncol. 2022 May 20;40(15):1671-1680. doi: 10.1200/JCO.21.02188. Epub 2022 Feb 18. PMID 35180010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 57 sites in 13 countries./territories.
Pre-assignment Details: Participants enrolled in Cohort 1a must have received ruxolitinib therapy for at least 12 weeks and currently be on a stable dose of ≥10 mg twice daily of ruxolitinib. For Cohort 1b, participants must have received prior treatment with ruxolitinib. For Cohort 2, participants must have received prior treatment with a JAK-2 inhibitor. For Cohort 3, participants must not have received prior treatment with a JAK-2 inhibitor or BET inhibitor.
Period: Overall Study
Arm/Group | Navitoclax + Ruxolitinib (Cohort 1a) | Navitoclax + Ruxolitinib (Cohort 1b) | Navitoclax (Cohort 2) | Navitoclax + Ruxolitinib (Cohort 3)
Started | 34 | 91 | 34 | 32
Completed | 0 | 0 | 0 | 0
Not Completed | 34 | 91 | 34 | 32
Not completed — Withdrew consent | 3 | 9 | 4 | 2
Not completed — Lost to Follow-up | 2 | 2 | 1 | 0
Not completed — Death | 20 | 38 | 18 | 10
Not completed — Other, not specified | 9 | 42 | 11 | 20

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who take at least one dose of navitoclax
Groups:
- Total: Total of all reporting groups
Arm/Group | Navitoclax + Ruxolitinib (Cohort 1a) | Navitoclax + Ruxolitinib (Cohort 1b) | Navitoclax (Cohort 2) | Navitoclax + Ruxolitinib (Cohort 3) | Total
Number analyzed (Participants) | 34 | 91 | 34 | 32 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (10.38) | 66.5 (9.26) | 69.0 (6.56) | 68.0 (10.10) | 67.4 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 34 | 14 | 12 | 71
  Male | 23 | 57 | 20 | 20 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 4 | 6 | 19
  Not Hispanic or Latino | 32 | 84 | 30 | 26 | 172
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 15 | 3 | 0 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 2 | 5
  White | 32 | 76 | 30 | 29 | 167
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥ 35% Reduction From Baseline in Spleen Volume at Week 24
Description: Reduction in spleen volume is measured by magnetic resonance imaging/computerized tomography (MRI/CT).
Time Frame: Baseline, Week 24
Population: Full Analysis Set (FAS): all participants who take at least one dose of navitoclax
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Navitoclax + Ruxolitinib (Cohort 1a) | Navitoclax + Ruxolitinib (Cohort 1b) | Navitoclax (Cohort 2) | Navitoclax + Ruxolitinib (Cohort 3)
Number analyzed (Participants) | 34 | 91 | 34 | 32
percentage of participants | 26.47 [12.88 to 44.36] | 21.98 [13.97 to 31.88] | 11.76 [3.30 to 27.45] | 62.50 [43.69 to 78.90]

2. Secondary Outcome: Percentage of Participants Achieving ≥ 50% Reduction From Baseline in Total System Score (TSS) at Week 24
Description: TSS is assessed by the Myelofibrosis Symptom Assessment Form (MFSAF) version 4.0. Participants complete a symptom diary and rate the following seven MF symptoms: fatigue, night sweats, abdominal discomfort, pruritus, pain under the ribs on the left side, early satiety, and bone pain daily using a scale from 0 (absent) to 10 (worst imaginable), and the scores are averaged over 7 days, with a minimum of 4 days required to calculate the average score. Participants for whom a valid average score cannot be calculated either at baseline or post-baseline are considered non-responders. The TSS reflects the sum of the scores of these symptoms, for a maximum possible score of 70 (i.e., most severe symptom experience).
Time Frame: Baseline, Week 24
Population: Full Analysis Set (FAS): all participants who take at least one dose of navitoclax
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Navitoclax + Ruxolitinib (Cohort 1a) | Navitoclax + Ruxolitinib (Cohort 1b) | Navitoclax (Cohort 2) | Navitoclax + Ruxolitinib (Cohort 3)
Number analyzed (Participants) | 34 | 91 | 34 | 32
percentage of participants | 20.59 [8.70 to 37.90] | 25.27 [16.75 to 35.47] | 8.82 [1.86 to 23.68] | 34.38 [18.57 to 53.19]

3. Secondary Outcome: Percentage of Participants Achieving Anemia Response
Description: For a participant who is transfusion independent (TI) at Baseline with hemoglobin value < 10 g/dL, anemia response is achieved if the post-Baseline hemoglobin level increases by ≥2 g/dL without receiving packed red blood cells (PRBC) transfusion (for any reason) within 2 weeks and without any erythropoietin or mimetics within the last 4 weeks prior to the increase in hemoglobin level by ≥2g/dL was observed. Hemoglobin values more than 30 days after the last dose of study treatment or after the start of post-study treatment or disease progression, whichever is earlier, will not be considered in the analysis of anemia response.
  For a participant who is transfusion dependent (TD) at Baseline, anemia response is defined as a period of at least 12 consecutive weeks without PRBC transfusion at any time after the first dose of study drug and on or prior to 30 days post last dose of study drug, the start of post-study treatment, disease progression or death, whichever occurs earlier.
Time Frame: Up to 254 weeks
Population: Full Analysis Set (FAS): all participants who take at least one dose of navitoclax; participants who were Baseline transfusion independent with baseline hemoglobin of ≥10 g/dL were excluded from the analysis since they were not evaluable for anemia response. Missing post-Baseline anemia response in Full Analysis Set applicable to evaluation of anemia response are considered as non-responders of anemia response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Navitoclax + Ruxolitinib (Cohort 1a) | Navitoclax + Ruxolitinib (Cohort 1b) | Navitoclax (Cohort 2) | Navitoclax + Ruxolitinib (Cohort 3)
Number analyzed (Participants) | 11 | 50 | 25 | 15
percentage of participants
  Baseline transfusion independent with Baseline HGB <10 g/dL: number analyzed (Participants) | 7 | 38 | 17 | 13
  Baseline transfusion independent with Baseline HGB <10 g/dL | 28.57 [3.67 to 70.96] | 23.68 [11.44 to 40.24] | 52.94 [27.81 to 77.02] | 38.46 [13.86 to 68.42]
  Baseline transfusion dependent: number analyzed (Participants) | 4 | 12 | 8 | 2
  Baseline transfusion dependent | 50.00 [6.76 to 93.24] | 16.67 [2.09 to 48.41] | 37.50 [8.52 to 75.51] | 100 [15.81 to 100.00]
  Overall | 36.36 [10.93 to 69.21] | 22.00 [11.53 to 35.96] | 48.00 [27.80 to 68.69] | 46.67 [21.27 to 73.41]

4. Secondary Outcome: Percentage of Participants With ≥ 1 Grade Reduction From Baseline in Fibrosis Grade At Any Time
Description: Bone marrow grading is assessed according to the European Consensus Grading System. The 4-point grading scale ranges from MF-0, which corresponds to normal bone marrow, to MF-3, diffuse and dense increase in reticulin with extensive intersections with coarse bundles of collagen, often associated with significant osteosclerosis.
Time Frame: Up to 254 weeks
Population: Full Analysis Set (FAS): all participants who take at least one dose of navitoclax; participants with missing bone marrow fibrosis grade (either Baseline or post-Baseline) or those with bone marrow fibrosis Grade 0 at Baseline were excluded from the analysis for the change in bone marrow fibrosis grade
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Navitoclax + Ruxolitinib (Cohort 1a) | Navitoclax + Ruxolitinib (Cohort 1b) | Navitoclax (Cohort 2) | Navitoclax + Ruxolitinib (Cohort 3)
Number analyzed (Participants) | 31 | 77 | 22 | 27
percentage of participants
  Week 24: number analyzed (Participants) | 26 | 54 | 15 | 23
  Week 24 | 23.08 [8.97 to 43.65] | 24.07 [13.49 to 37.64] | 40.00 [16.34 to 67.71] | 30.43 [13.21 to 52.92]
  Anytime during the post-Baseline period | 41.94 [24.55 to 60.92] | 41.56 [30.43 to 53.36] | 40.91 [20.71 to 63.65] | 48.15 [28.67 to 68.05]

5. Secondary Outcome: Time to First Reduction in Fibrosis Grade
Description: Grade of bone marrow fibrosis was assessed by investigators according to the European Consensus Grading System. The 4-point grading scale ranges from MF-0, which corresponds to normal bone marrow, to MF-3, diffuse and dense increase in reticulin with extensive intersections with coarse bundles of collagen, often associated with significant osteosclerosis. The time to first achieving a reduction of at least 1 grade in bone marrow fibrosis from Baseline was summarized.
Time Frame: Up to 254 weeks
Population: Full Analysis Set (FAS): all participants who take at least one dose of navitoclax; participants with Baseline bone marrow fibrosis grade >0 and post-Baseline bone marrow fibrosis grade are included in the analysis
Measure: Median (Full Range); unit: weeks
Arm/Group | Navitoclax + Ruxolitinib (Cohort 1a) | Navitoclax + Ruxolitinib (Cohort 1b) | Navitoclax (Cohort 2) | Navitoclax + Ruxolitinib (Cohort 3)
Number analyzed (Participants) | 13 | 32 | 9 | 13
weeks | 24.1 [11.1 to 107.1] | 24.1 [9.3 to 97.1] | 12.4 [11.9 to 48.1] | 12.3 [7.0 to 96.1]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events tables include events reported from the time of informed consent to the end of the study. Median time on follow-up was for 76.1 months for Navitoclax + ruxolitinib (Cohort 1a); 41.9 months for Navitoclax + ruxolitinib (Cohort 1b); 40.2 months for Navitoclax (Cohort 2); and 44.2 months for Navitoclax + ruxolitinib (Cohort 3).
Groups:
- Navitoclax + Ruxolitinib (Cohort 1b): Those receiving ruxolitinib at Screening must be on a stable dose ≥10 mg tablets orally twice daily (BID) for ≥4 weeks prior to 1st dose of navitoclax. Those not receiving ruxolitinib at Screening received 10 mg ruxolitinib BID starting on Day 1. Navitoclax tablets were administered orally once daily (QD) per Baseline platelet count (>150 × 10^9/L starting dose of 200 mg; ≤150 × 10^9/L starting dose of 100 mg, which could be increased to 200 mg QD after 7 days provided platelet count is ≥75 × 10^9/L). Navitoclax didn't exceed 200 mg QD for first 24 weeks of treatment. After Week 24 disease assessment, navitoclax dose was increased to 300 mg QD at discretion of the Investigator for those with suboptimal spleen response defined as failure to achieve spleen volume reduction of at least 10% per imaging. Participants continued their treatment until the end of clinical benefit, unacceptable toxicity, or they met other protocol criteria for discontinuation (whichever occurred first).
Arm/Group | Navitoclax + Ruxolitinib (Cohort 1a) | Navitoclax + Ruxolitinib (Cohort 1b) | Navitoclax (Cohort 2) | Navitoclax + Ruxolitinib (Cohort 3)
All-Cause Mortality (participants affected / at risk) | 20/34 | 39/91 | 18/34 | 10/32
Serious Adverse Events (participants affected / at risk) | 21/34 | 35/91 | 18/34 | 12/32
Other Adverse Events (participants affected / at risk) | 34/34 | 91/91 | 34/34 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navitoclax + Ruxolitinib (Cohort 1a) (N=34) | Navitoclax + Ruxolitinib (Cohort 1b) (N=91) | Navitoclax (Cohort 2) (N=34) | Navitoclax + Ruxolitinib (Cohort 3) (N=32)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIAC DISORDER (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRIC VARICES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL ANGIODYSPLASIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRUG WITHDRAWAL SYNDROME (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GENERALISED OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 2 (3) | 1 (3) | 0 (0) | 1 (1)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANORECTAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 4 (5) | 2 (2) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENTEROBACTER SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GIARDIASIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
IMPLANT SITE CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYCOBACTERIAL INFECTION (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
ORAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 6 (9) | 2 (3) | 0 (0) | 0 (0)
PNEUMONIA MORAXELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
VARICELLA ZOSTER VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IMMUNISATION REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LISFRANC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TROPONIN I INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUROENDOCRINE CARCINOMA OF THE SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL CELL CARCINOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
TRANSFORMATION TO ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
DEMENTIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTRACRANIAL HAEMATOMA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PELVIC HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EMBOLISM (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
VASCULITIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navitoclax + Ruxolitinib (Cohort 1a) (N=34) | Navitoclax + Ruxolitinib (Cohort 1b) (N=91) | Navitoclax (Cohort 2) (N=34) | Navitoclax + Ruxolitinib (Cohort 3) (N=32)
ANAEMIA (Blood and lymphatic system disorders) | 11 (23) | 47 (81) | 13 (26) | 21 (51)
EOSINOPHILIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
LEUKOPENIA (Blood and lymphatic system disorders) | 2 (8) | 5 (7) | 1 (1) | 1 (4)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 1 (1) | 3 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (8) | 13 (28) | 6 (15) | 10 (20)
SPLENOMEGALY (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 30 (134) | 45 (146) | 10 (28) | 18 (75)
EAR PAIN (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
VISION BLURRED (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
VITREOUS FLOATERS (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 3 (3) | 5 (6) | 1 (1) | 4 (5)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 5 (5) | 4 (6) | 5 (5) | 3 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 (8) | 11 (16) | 5 (6) | 6 (10)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 7 (8) | 4 (6) | 1 (1) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 5 (5) | 10 (13) | 3 (4) | 5 (7)
DIARRHOEA (Gastrointestinal disorders) | 27 (51) | 47 (76) | 15 (27) | 18 (45)
DYSPEPSIA (Gastrointestinal disorders) | 3 (5) | 6 (6) | 3 (3) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 4 (4) | 2 (3) | 2 (2) | 3 (4)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (3)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
MOUTH ULCERATION (Gastrointestinal disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 15 (19) | 26 (30) | 12 (19) | 10 (16)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 8 (9) | 1 (1) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 7 (9) | 6 (6) | 5 (8) | 4 (5)
ASTHENIA (General disorders) | 0 (0) | 8 (9) | 2 (3) | 3 (4)
CHILLS (General disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
EARLY SATIETY (General disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 24 (38) | 17 (23) | 9 (11) | 9 (9)
INFLUENZA LIKE ILLNESS (General disorders) | 3 (4) | 2 (2) | 0 (0) | 1 (2)
OEDEMA (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 6 (7) | 11 (15) | 5 (6) | 3 (4)
PAIN (General disorders) | 1 (1) | 6 (6) | 1 (1) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 3 (3) | 1 (1) | 2 (3) | 0 (0)
PYREXIA (General disorders) | 3 (3) | 9 (14) | 3 (3) | 3 (4)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 3 (3) | 8 (12) | 2 (2) | 2 (2)
JAUNDICE (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 5 (6) | 22 (23) | 8 (10) | 12 (15)
EAR INFECTION (Infections and infestations) | 3 (5) | 3 (3) | 0 (0) | 0 (0)
FOLLICULITIS (Infections and infestations) | 2 (2) | 3 (4) | 1 (1) | 0 (0)
GENITAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
HERPES ZOSTER (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
ORAL HERPES (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
PHARYNGITIS (Infections and infestations) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
RHINITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 3 (4) | 2 (2) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 (16) | 6 (7) | 4 (4) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 6 (10) | 7 (14) | 4 (4) | 4 (4)
CONTUSION (Injury, poisoning and procedural complications) | 13 (16) | 9 (11) | 2 (2) | 3 (4)
FALL (Injury, poisoning and procedural complications) | 6 (7) | 2 (2) | 6 (8) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 8 (10) | 9 (15) | 4 (5) | 7 (12)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 6 (9) | 11 (16) | 6 (7) | 7 (11)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 5 (9) | 6 (7) | 3 (5) | 3 (5)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (8) | 12 (15) | 7 (8) | 5 (9)
BLOOD CREATININE INCREASED (Investigations) | 5 (5) | 5 (5) | 3 (3) | 1 (1)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 5 (5) | 2 (2) | 3 (4)
C-REACTIVE PROTEIN INCREASED (Investigations) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
CARDIAC MURMUR (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
EASTERN COOPERATIVE ONCOLOGY GROUP PERFORMANCE STATUS WORSENED (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3 (7) | 2 (3) | 0 (0) | 2 (2)
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 (3) | 9 (29) | 2 (2) | 6 (20)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (4) | 17 (49) | 6 (19) | 5 (9)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 37 (103) | 10 (20) | 12 (36)
WEIGHT DECREASED (Investigations) | 3 (4) | 8 (11) | 5 (5) | 1 (1)
WEIGHT INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 3 (6) | 15 (39) | 4 (8) | 6 (14)
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 (7) | 9 (11) | 6 (7) | 1 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
FOLATE DEFICIENCY (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (9)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 4 (5) | 2 (2) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 (2) | 3 (6) | 1 (1) | 2 (2)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 6 (7) | 14 (17) | 5 (7) | 4 (4)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (6) | 1 (1) | 3 (3)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 (2) | 9 (19) | 5 (5) | 4 (8)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 (2) | 4 (6) | 2 (2) | 6 (9)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 3 (6) | 3 (3) | 3 (7)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 10 (14) | 11 (14) | 5 (5) | 5 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (5) | 2 (2) | 3 (3)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (2)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (6) | 3 (3) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1) | 0 (0) | 4 (5)
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 10 (13) | 11 (13) | 4 (4) | 6 (6)
HEADACHE (Nervous system disorders) | 7 (7) | 12 (12) | 4 (5) | 4 (7)
PARAESTHESIA (Nervous system disorders) | 3 (3) | 5 (5) | 0 (0) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (3)
TASTE DISORDER (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
INSOMNIA (Psychiatric disorders) | 4 (6) | 6 (6) | 3 (3) | 2 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 8 (9) | 3 (3) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 3 (4) | 4 (5) | 3 (3)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 8 (8) | 1 (1) | 3 (3)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
AQUAGENIC PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (3) | 2 (2) | 1 (1)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (9) | 1 (1) | 2 (2)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (4) | 13 (15) | 5 (6) | 6 (8)
RASH (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (4) | 2 (2) | 4 (4)
SKIN LESION (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3) | 0 (0) | 4 (5)
HAEMATOMA (Vascular disorders) | 2 (2) | 1 (5) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 3 (5) | 8 (8) | 2 (2) | 3 (3)
HYPOTENSION (Vascular disorders) | 2 (3) | 2 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT03222609/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT03222609/SAP_001.pdf